CLINICAL TRIAL: NCT07095569
Title: Shoulder Denervation as Management of Post Mastectomy Irradiation Shoulder Pain: Randomized Control Trial
Brief Title: Shoulder Denervation for Post Mastectomy Irradiation Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Suzan Adlan Abdelrahman, Assistant professor, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IORG003381
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Shoulder individual nerves TRF (thermal radio frequency): Patients will receive shoulder i (Experimental): Thermal RF therapy will be performed under ultrasound guidance.
  Interventions: Device: (Shoulder individual nerves TRF (thermal radio frequency): Patients will receive shoulder individual nerves Thermal RF.
- Group 2 (Control): Patients will receive conservative treatment. (Active Comparator): Patients will receive conservative treatment Acetaminophen (paracetamol) 1000 mg tid and pregabalin (lyrica)75 mg bid; can be increased to 150 mg bid, oxycodone (oxynorm) 10mg IR PRN.
  Interventions: Drug: conservative treatment

INTERVENTIONS:
Device: (Shoulder individual nerves TRF (thermal radio frequency): Patients will receive shoulder individual nerves Thermal RF. — Shoulder individual nerves thermal RF technique: The patient will be put in the sitting position, monitored with electrocardiography, pulse oximetry, and non-invasive blood pressure. after disinfection A high-frequency linear transducer (10-15 Hz) will be placed parallel and cephalad to the spine of the scapula. The probe will be moved from cephalad to caudad until the trapezius and supraspinatus muscles were identified. The suprascapular nerve will be identified as a hyperechogenic structure in the suprascapular fossa deep to the superior transverse scapular ligament. A 10 cm radiofrequency needle, with a 10 mm active tip, will be inserted in plane with the ultrasound beam and advanced to reach the proximity to the nerve. A nerve stimulator was used as an additional nerve-finding modality.
  Arms: Group 1 (Shoulder individual nerves TRF (thermal radio frequency): Patients will receive shoulder i
Drug: conservative treatment — Patients will receive conservative treatment Acetaminophen (paracetamol 1000 mg tid and pregabalin (lyrica) 75 mg bid; can be increased to 150 mg bid, oxycodone (oxynorm) 10mg IR PRN.
  Arms: Group 2 (Control): Patients will receive conservative treatment.

SUMMARY:
Breast cancer is the second most common cancer world-wide following lung cancer. It afflicts about 1.7 million patients annually, of which 60% mandate surgery of the breast and/or the axilla, and nearly 20-50% of them may develop post mastectomy pain syndrome .

After breast cancer surgery, between 6% and 86% of people may develop tight bands of fibrous tissue under their skin, known as axillary web syndrome. These bands can cause pain in the shoulder area by trying to raise or extend the arm. Shoulder pain is a common side effect of breast cancer surgery and treatment.

Various medical and interventional procedures have been tried for treating postmastectomy shoulder pain, with varying efficacy . Among the interventional procedures that may have a role for treatment.

Innervation of the glenohumeral joint (GHJ) can be divided into anterior and posterior innervation from articular branches of the suprascapular nerve (SN):C5 &6 (posterior-lateral), axillary nerve (AN):C5 &6 (anterior-lateral, inferior, and posteriorlateral), and lateral pectoral nerve (LPN): C5 &6 (anterior superior)

DETAILED DESCRIPTION:
The investigators hypothesize that thermal RF (radiofrequency) of shoulder individual nerves is efficacious for the management of post-mastectomy shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age (18-65) Years.
2. ASA physical status (II- III).
3. Patients with post mastectomy irradiation shoulder pain.
4. Body mass index (BMI): (20-40) kg/m2.

Exclusion Criteria:

1. Patient refusal.
2. Known sensitivity or contraindication to drugs used in the study.
3. Pregnancy.
4. Recent myocardial infarction.
5. Hemodynamically unstable.
6. Local and systemic sepsis.
7. Psychiatric illness.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Assess the changes in NPRS (numerical pain rating scale) for assessment of pain relief which will be recorded before treatment and at 1 month, 2 months and 3-month intervals following treatment. | 1 month, 2 months and 3-month intervals following treatment.
  numerical pain rating scale is a measurement tool that uses numbers to represent the intensity of a characteristic or quality, where 0 might represent "no pain" and 100 the highest number represents "the worst pain imaginable".

SECONDARY OUTCOMES:
Measure oxycodone IR (immediate release) consumption | 1 month, 2 months and 3-month intervals following treatment.

IPD SHARING:
Plan to Share IPD: Undecided